CLINICAL TRIAL: NCT06171347
Title: The Effect of Oral Cold Water Spray Application on Thirst Severity in Patients Undergoing Spinal Surgery: A Randomised Controlled Trial
Brief Title: The Effect of Oral Cold Water Spray Application on Thirst Severity in Patients Undergoing Spinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Zeynep Kızılcık Ozkan, Assistant professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/349
Record Dates: First submitted 2023-11-27; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Thirst

STUDY DESIGN:
Intervention Model Description: Patients in the experimental group will receive oral cold spray in the postoperative period.
  Patients in the control group will receive standard care in the postoperative period.
Who Masked: Outcomes Assessor
Masking Description: The data will be collected and coded by the nurse researcher. Data will be analyzed by an independent statistician. The study groups will be disguised as A and B. The statistician will not know the groups. In addition, the statistical expert will not see the data of the experimental group regarding satisfaction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients in the experimental group will receive oral cold spray (tap water) in the postoperative period.
  Interventions: Other: Oral cold spray (tap water)
- Control group (No Intervention): Patients in the control group will not be intervened in the postoperative period except for standard care for thirst management.

INTERVENTIONS:
Other: Oral cold spray (tap water) — Oral cold spray (tap water)
  Arms: Experimental group

SUMMARY:
The aim of this study was to determine the effect of oral cold water spray application on thirst severity and patient satisfaction after spinal surgery.

H1: Oral cold water spray application has an effect on thirst severity after spinal surgery.

H2: Oral cold water spray application has an effect on salivary pH after spinal surgery.

H3: Oral cold water spray application affects the satisfaction of patients after spinal surgery.

DETAILED DESCRIPTION:
The randomized controlled trial will be conducted in the brain and neurosurgery service of Trakya University Health Research and Application Centre. Date of research will be conducted between December 2023 and March 2024. The research sample will consist of 62 volunteer patients. The sample was determined using power analysis at the research planning stage. The minimum number of people to be included in the sample was calculated as 62, each group consisting of 31 (1:1) patients, with an effect size of 0.75, 95% confidence level, 5% tolerance and 80% power ratio, using the G.Power 3.1.9.4 program. Data Collection Forms Patient information form; The form was developed by the researchers in line with the literature and consisted of 9 questions inquiring information about age, gender, educational status, height, body weight, marital status, habits, physician diagnosis, presence of chronic diseases, etc.

ostoperative patient follow-up form; There are 11 questions in the form. The answers to the first 9 questions will be obtained by interviewing the patient face to face. The eleventh question (type of fluid taken during surgery) and the answer to the twelfth question (amount of bleeding during surgery) will be obtained from the anaesthesia transfer form.

The severity of thirst and discomfort levels of the patients will be evaluated numerically four times and saliva pH levels will be evaluated twice (before the first application and 1 hour after the end of the whole application) with the chart at the end of the form (Visual Analogue Scale values). The Visual Analogue Scale, which is used to convert data that cannot be evaluated numerically into numerical form, is 10 cm long and is graded on a horizontal or vertical line. Since thirst is a state of discomfort consisting of subjective experiences expressed by the person, it is stated in the literature that the use of the Visual Analogue Scale in the evaluation of thirst is appropriate and can be used safely in studies. The scale includes 2 questions evaluating the severity of thirst and the severity of discomfort from thirst numerically between 0-10. Patient satisfaction form; The satisfaction of the patients in the experimental group with the oral cold water spray application will be evaluated with a numerical rating scale ranging from 0 to 10 points (0 = I am not satisfied at all, 10 = I am very satisfied).

Data collection process Patients who meet the inclusion criteria will be informed verbally and in writing about the study, scales, etc. in the preoperative period and the informed consent form will be signed. "Patient Information Form" will be applied in the preoperative period. The data of the study will be collected by the researcher in the patient room by face-to-face interview method.

On postoperative day 0, all patients will be verbally informed by the ward nurses about the standard guidelines and care to be followed after spinal surgery after admission to the ward.

Patients in the control group will not receive any intervention to quench thirst. The questions in the postoperative patient follow-up form will be asked by the researcher and the postoperative patient follow-up form will be filled out.

After the standard care of the service is applied to the patients in the experimental group, the patients will be evaluated by the researcher nurse with the "Safe Protocol in the Management of Thirst in the Early Postoperative Period" in the 2nd postoperative hour after admission to the service. The postoperative patient follow-up form will be applied to patients with appropriate criteria. Saliva pH will be evaluated before the first set. Afterwards, 0.5 ml of oral cold water spray kept in the 40C service refrigerator will be applied. Thirty minutes later, 0.5 ml of oral cold water spray which has been kept in the 40C service refrigerator will be applied for the second time. The first set will be completed. In the third hour, the severity of thirst and discomfort due to thirst will be evaluated with the chart in the postoperative patient follow-up form. In the fourth hour, 0.5 ml oral cold water spray kept in the 40C service refrigerator will be applied. Thirty minutes later, 0.5 ml of oral cold water spray kept in the 40C service refrigerator will be applied again. The second set will be completed. In the fifth hour, the severity of thirst and discomfort due to thirst and saliva Ph will be evaluated with the chart in the postoperative patient follow-up form. In addition, patients' satisfaction with oral cold water spray application will be evaluated. Data collection will end after the completion of the questionnaire applications.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient treatment in the neurosurgery ward,
* undergoing planned spinal surgery under general anaesthesia,
* Admitted to the ward after surgery,
* Who volunteered to participate in the research,
* No mental disability,
* 18 years of age,
* Literate,
* Accepting random selection,
* Patients without communication problems in Turkish

Exclusion Criteria:

* Spinal surgery performed under spinal anaesthesia,
* Admitted to intensive care or external ward after surgery,
* Emergency surgery,
* not volunteering to participate in the research,
* Mentally handicapped,
* Under 18 years of age,
* Illiterate,
* which does not accept random selection,
* Patients with communication problems in Turkish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
thirst | postoperative period (2., 2.5, 4. and 4.5. hours)
  to determine the effect of oral cold water spray application on the severity of thirst after spinal surgery.
  Thirst severity and discomfort levels of the patients will be evaluated numerically four times and salivary pH levels will be evaluated twice (before the first application and 1 hour after the end of all applications) with the chart (Visual Analogue Scale values) at the end of the "Postoperative patient follow-up form". The Visual Analogue Scale, which is used to convert data that cannot be evaluated numerically into numerical form, is 10 cm long and is graded on a horizontal or vertical line. Since thirst is a state of discomfort consisting of subjective experiences expressed by the person, it is stated in the literature that the use of the Visual Analogue Scale in the evaluation of thirst is appropriate and can be used safely in studies.

SECONDARY OUTCOMES:
satisfaction of patients | postoperative period (6.hour)
  to determine the effect of oral cold water spray application on patient satisfaction after spinal surgery.
  Patient satisfaction form; The satisfaction of the patients in the experimental group with the oral cold water spray application will be evaluated with a numerical rating scale ranging from 0 to 10 points (0 = I am not satisfied at all, 10 = I am very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Turkey, Trakya University, Edirne, Turkey (Türkiye)